CLINICAL TRIAL: NCT07372183
Title: Wound Healing Following Extraction and Ridge Preservation in Smokers and Non-smokers
Status: Not yet recruiting | Type: Observational
Sponsor: Marquette University (Other)
Collaborators: LifeNet Health (Industry)
Responsible Party: Principal Investigator, Vrisiis Kofina, Director, Advanced Education in Periodontics Program, Assistant Professor of Periodontics, Marquette University
Other Study IDs: HR-4728
Record Dates: First submitted 2025-12-02; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Smoking, Cigarette; Alveolar Bone Grafting; Wound Healing; Bone Healing; Tooth Extraction Site Healing
MeSH Terms: conditions — Cigarette Smoking | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bone cores will be harvested at the time of implant placement using trephine drills via surgical guides.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Smokers: Subjects are qualified as smokers if they report smoking ≥10 cigarettes/day for ≥5 years, and maintain a 8ppm carbon monoxide concentration or higher via smokerlyzer test.
  Interventions: Other: observational study
- Non-smokers: Subjects qualify as nonsmokers if they have never smoked and upon confirmation by the smokerlyzer test of carbon monoxide concentation of less than 8ppm.
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — Observational study; alveolar ridge preservation

SUMMARY:
The goal of this study is to evaluate bone wound healing following extraction and alveolar ridge preservation (bone graft and membrane) clinically, histologically and in relation to gene expression in smokers and non-smokers. Data from a small group of participants will be analyzed after age-matched subjects undergo extraction and alveolar ridge preservation prior to implant placement. The data obtained in this pilot study will be used to plan a full-fledged study involving a larger number of smoking and non-smoking participants to compare the two groups.

DETAILED DESCRIPTION:
All research procedures will start after IRB approval. Patients of the Graduate Periodontics Clinic in need of extraction, bone graft and membrane will be recruited. There will be two groups (smokers and non-smokers) and their demographic and social, periodontal, surgery-related, anatomical and healing variables as well as patient-reported outcomes will be recorded at different time points (immediately before, during and immediately after surgery and 1, 2, 6 weeks and 4 months) in order to evaluate wound healing outcomes and differences between the groups. The demographic and social variables evaluated are age, gender, race, medical history, medications, smoking (via interview and breath test-smokerlyzer) and alcohol consumption (via interview). The periodontal variables are tooth mobility, probing depth, attachment level, gingival and plaque index. The surgery-related variables include intraoperative complications, duration of procedure, anesthetic amount, type and approach and operator experience. The anatomical variables are bone height and width (buccolingual and buccal dimension), bone density (in Cone Beam Computed Tomographies - CBCTs) and gingival width and thickness. The healing variables include wound opening (tested clinically and in photos), bleeding, grafting material discharge, flap necrosis, loose sutures, and temporary restoration adjustment. The patient-reported outcomes are Oral Health Impact Questionnaire-14 (OHIP-14), Visual Analogue Scale (VAS) for pain, swelling and difficulty of mouth opening. At 4 months during the implant placement appointment, a bone core will be harvested via a 3D printed surgical guide based on virtual CBCT planning. The core willl be used of microCT and histological analysis as well as total RNA extraction and RNA sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18-75 years)
* Good general health (controlled conditions)
* Smokers (≥10 cigarettes/day for ≥5 years) and never smokers. Confirmation of smoking status will be done via use of a smokerlyzer. The cut-off point for distinguishing smokers from non-smokers is 8 carbon monoxide parts per million (ppm).
* Periodontal status: periodontal health, gingivitis on intact or reduced periodontium, treated periodontitis
* Intact post-extraction bony walls or less than 50% bone dehiscence
* Distance at least 8 mm of vertical bone height between bone crest and anatomical structures (i.e. sinus floor, inferior alveolar nerve (IAN) canal, mental foramen)
* Extracted tooth root in the same three-dimensional position as the future implant placement so that the bone core biopsy can be taken from a site totally within the confines of the former tooth socket without inclusion of surrounding native alveolar bone
* Scheduled for single tooth extraction with bone graft placement and membrane

Exclusion Criteria:

* Uncontrolled periodontal disease
* Uncontrolled systemic disease
* Pregnancy
* Use of therapy and/or medication that impairs wound healing (e.g., bisphosphonates, steroids, chemotherapy, radiotherapy etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for tooth extraction and alveolar ridge preservation (bone graft and membrane) in the Graduate Periodontics Clinic at Marquette University School of Dentistry.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2026-01-25 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Parameters | Measured before surgery, during surgery and at 4 months
  bone width
Clinical Parameters | Measured before surgery, during surgery and at 4 months
  bone height

SECONDARY OUTCOMES:
Genetic Parameters | Bone samples harvested at 4 months
  RNA transcriptomic analysis
Histological Parameters | Samples harvested at 4 months
  Histological analysis of bone cores: %mineralized bone
Histological Parameters | Samples harvested at 4 months
  Histological analysis of bone cores: %osteoid
Histological Parameters | Samples harvested at 4 months
  Histological analysis of bone cores: %residual bone graft
Histological Parameters | Samples harvested at 4 months
  Histological analysis of bone cores: %soft tissue
Histological Parameters | Samples harvested at 4 months
  Histological analysis of bone cores: numbers of osteoblasts and osteoclasts
Micro-CT Parameters | Samples harvested at 4 months
  Histological analysis of bone cores: bone mineral density
Micro-CT Parameters | Samples harvested at 4 months
  Histological analysis of bone cores: tissue mineral density
Micro-CT Parameters | Samples harvested at 4 months
  Histological analysis of bone cores: bone volume / tissue volume (BV/TV)
Micro-CT Parameters | Samples harvested at 4 months
  Histological analysis of bone cores: trabecular number
Micro-CT Parameters | Samples harvested at 4 months
  Histological analysis of bone cores: trabecular separation
Micro-CT Parameters | Samples harvested at 4 months
  Histological analysis of bone cores: trabecular thickness
Patient-reported Parameters | Measured before surgery, at 1, 2 and 6 weeks, and 4 months
  Oral Health Impact Profile -14 (OHIP-14). Range from 0 (no impact) to 56 (most severe impact).
Patient-reported Parameters | Measured before surgery and at 1, 2 and 6 weeks, and 4 months
  VAS for pain (0-100). Zero indicates no pain and 100 the worst pain imaginable.
Patient-reported Parameters | Measured before surgery and at 1, 2 and 6 weeks, and 4 months
  VAS for swelling (0-100). Zero indicates no swelling and 100 the worst swelling imaginable.
Patient-reported Parameters | Measured before surgery, at 1, 2 and 6 weeks, and 4 months
  VAS for difficulty of mouth opening (0-100). Zero indicates no difficulty of mouth opening and 100 complete inability to open mouth.

OTHER OUTCOMES:
Clinical Parameters | Measured at baseline (before surgery)
  gingival width
Clinical Parameters | Measured at baseline (before surgery)
  gingival thickness
Clinical Parameters | Measured immediately after surgery, at 1, 2 and 6 weeks and 4 months
  wound opening
Clinical Parameters | Measured at 1, 2 and 6 weeks and 4 months
  bleeding
Clinical Parameters | Measured at 1, 2 and 6 weeks and 4 months
  grafting material discharge
Clinical Parameters | Measured at 1, 2 and 6 weeks and 4 months
  flap necrosis

CONTACTS AND LOCATIONS:
Overall Officials: Vrisiis Kofina, DDS, MS, Principal Investigator — Marquette University
Locations (1):
- Marquette University School of Dentistry Graduate Periodontics Clinic, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No